CLINICAL TRIAL: NCT05346939
Title: To Analyze the Kinematic Change of Lower Limb During Jumping Task With Wearable Device - 2-year Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202101717B0
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-04

CONDITIONS: Landing Error Scoring System (LESS)
Keywords: Dynamic taping; Landing Error Scoring System (LESS); ACL injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: The first year, the investigators would verify the relation between wearable device and motion analysis and its validity and reliability (n=15). And the investigators are going to observe the effect of dynamic taping in lower limb biomechanics of high-school soccer and basketball athletes (n=50). In the second year, the investigators would recruit high school soccer and basketball athletes to examine the effect of dynamic taping in lower limb biomechanics under fatigue (n=50). In order to exclude the influence of sequence and learning effect, a cross-over study was used, and the interval between the two tests was about 2 weeks.
Masking Description: In this study, the athletic trainer will intervene with a dynamic tape (spiral dynamic technique) using a dynamic tape for the first test and a sham dynamic tape for the second test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Senior high school athletes in Taiwan (Experimental): In the first year, the investigators would verify the relation between wearable device and motion analysis and its validity and reliability at stage I (n=15). And the investigators are going to observe the effect of dynamic taping in lower limb biomechanics of high-school soccer or basketball athletes (n=50) at stage II.
  In the second year, the investigators would recruit high school soccer and basketball athletes to examine the effect of dynamic taping in lower limb biomechanics under fatigue (n=50).
  Interventions: Device: dynamic taping

INTERVENTIONS:
Device: dynamic taping — The athletic trainer will intervene with spiral dynamic technique by using a dynamic tape for the first test and a sham dynamic tape for the second test, or reverse the order.

SUMMARY:
This study will be conducted in two years: In the first year, the investigators would verify the relation between wearable device and motion analysis and its validity and reliability. In advance, the investigators are going to observe the effect of dynamic taping in lower limb biomechanics of high-school soccer and basketball athletes. In the second year, the investigators would recruit high school soccer and basketball athletes to examine the effect of dynamic taping in lower limb biomechanics under fatigue.

DETAILED DESCRIPTION:
In Taiwan, it was estimated that at least 1,000 cases of patients require anterior cruciate ligament (ACL) reconstruction annually. Despite the improving of surgical technique, there are only 65% patients who received the ACL reconstruction return to their pre-injury level of sport. Therefore, to prevent ACL injuries in athletes is critical. The mechanism of ACL injury is greatly associated with lower limb biomechanics.

Motional analysis is the golden standard for biomechanics. However, with the advancement in technology, the investigators could explore lower limb biomechanics conveniently by wearable device. But the validity and reliability need further confirmation.

According to previous studies, the investigators could predict the possibility of ACL injuries by the change of biomechanics, such as hip adduction, internal rotation and knee valgus. Dynamic taping is a newly developing technique with better elasticity and extensibility. Studies showed that dynamic taping improve the biomechanics of knee joint. Hence, the investigators can adjust the faulty movement as soon as possible to prevent the occurrence of ACL injuries.

This study will be conducted in two years: In the first year, the investigators would verify the relation between wearable device and motion analysis and its validity and reliability. In advance, the investigators are going to observe the effect of dynamic taping in lower limb biomechanics of high-school soccer and basketball athletes. In the second year, the investigators would recruit high school soccer and basketball athletes to examine the effect of dynamic taping in lower limb biomechanics under fatigue.

ELIGIBILITY:
Inclusion Criteria:

* 1st Year: 16+ health volunteers
* 2nd Year: senior high school and college athlete

Exclusion Criteria:

* Those who are unable to exercise due to acute joint, muscle or nerve injury in the lower extremities
* Lower extremity surgery within 1 year
* Head trauma within 6 months
* Those with vestibular injury within 6 months
* Allergic to Dynamic tape
* Pregnant
* Visual coordination impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Understand the correlation between wearable devices (KinMAS system) and Vicon dynamic analysis system, and further assessment of the reliability and validity of the wearable devices (KinMAS system). | 1st Year
  The investigators would recruit health volunteers (n=15) to verify the relation between wearable device and motion analysis and its validity and reliability. Vicon motion capture system (golden standard) and wearable device (KinMAS system) are used simultaneously to measure the angle changes of the trunk and lower limbs with jump-landing task and counter movement jump.
Observe the effect of dynamic taping in lower limb biomechanics. | 1st Year
  The investigators would recruit senior high school athletes (n=50) to compare the changes of trunk and lower extremities joint angles with dynamic taping intervention. Subjects need to wear the wearable device (KinMAS system) and take double-leg Landing Error Scoring System (LESS) Score test with dynamic taping intervention. The athletic trainer will intervene with spiral dynamic technique by using a dynamic tape for the first test and a sham dynamic tape for the second test, or reverse the order. The Landing Error Scoring System (LESS) with double-leg consists of 17 items; total score is 0-19 points. Higher scores mean a worse outcome.
Observe the effect of dynamic taping in lower limb biomechanics after fatigue protocol. | 2nd Year
  The investigators would recruit senior high school athletes (n=50) to compare the changes of trunk and lower extremities joint angles with dynamic taping intervention. Subjects need to wear the wearable device (KinMAS system) and take double-leg and single-leg Landing Error Scoring System (LESS) Score tests with dynamic taping intervention after fatigue protocol. The athletic trainer will intervene with spiral dynamic technique by using a dynamic tape for the first test and a sham dynamic tape for the second test, or reverse the order. The Landing Error Scoring System (LESS) with double-leg consists of 17 items, total score is 0-19 points, whereas the single-leg consists of 14 items and total score is 0-16 points. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: CHIEN-HUNG CHEN, MD, Principal Investigator — Taoyuan Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No